CLINICAL TRIAL: NCT03147313
Title: Extracorporal Shock Wave Treatment After Microsurgical Coaptation to Improve Nerve Regeneration
Brief Title: Extracorporal Shock Wave Treatment to Improve Nerve Regeneration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ludwig Boltzmann Gesellschaft (Other)
Responsible Party: Principal Investigator, Rudolf Rosenauer, Principal investigator, Ludwig Boltzmann Gesellschaft
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MPG 07/2016
Record Dates: First submitted 2017-04-21; First posted 2017-05-10 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Peripheral Nerve Injury
Keywords: extracorporeal shock wave; microsurgical nerve coaptation; nerve regeneration
MeSH Terms: conditions — Peripheral Nerve Injuries

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into three groups: Two treatment groups with different treatment settings and one sham group.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant will be wearing an acoustic and visual masking. The outcome assessor won't know if the participant was treated or if he was assigned to the sham group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sham (Sham Comparator)
  Interventions: Device: Sham
- Shockwave 300 pulses (Active Comparator): 300 pulses of extracorporeal shock wave will be applied
  Interventions: Device: MTS Medical UG Orthogold 100
- Shockwave 500 pulses (Active Comparator): 500 pulses of extracorporeal shock wave will be applied
  Interventions: Device: MTS Medical UG Orthogold 100

INTERVENTIONS:
Device: MTS Medical UG Orthogold 100 — 300 or 500 pulses, frequency 3Hz, energy 1 (0,1mJ/mm2)
  Arms: Shockwave 300 pulses; Shockwave 500 pulses
Device: Sham — Extracorporeal shock wave treatment will be faked.
  Arms: Sham

SUMMARY:
This study evaluates the impact of extracorporeal shock wave treatment after microsurgical coaptation of finger nerves. Participants will be randomized into two treatment groups with different settings and a sham group. The participants will thereafter followed-up in a prospective, double-blind study design.

DETAILED DESCRIPTION:
Extracorporeal shock wave treatment is CE certified in Austria, Europe and licensed for indications like achillodynia, epicondylitis, or tendinitis calcanea. The Orthogold 100 device by MTS Medical UG will be used for this study.

Defocused low-energy extracorporeal shock wave therapy (ESWT) has gained acceptance as a therapeutic tool in different medical settings. It has been shown, that shock waves stimulate of the metabolic activity of different cell type, including osteoblasts, tenocytes, endothelial cells and chondrocytes. Furthermore, it has proved effective in clinical applications relating to bone and wound healing and myocardial ischaemia. Until now, no studies have been performed regarding the effects of ESWT on regeneration of peripheral nerve injuries in humans.

ELIGIBILITY:
Inclusion Criteria:

* complete lossless transection of one or more digital nerves distal to the branching out of the commune median or ulnar nerves
* direct, tension-free coaptation of the nerve stumps

Exclusion Criteria:

* segment loss of the nerve
* tension after direct coaptation
* diabetic neuropathy or other peripheral neuropathies
* other disease with reduced sensibility of the fingers
* injuries in the course of the nerve (plexus brachialis, median or ulnar nerve)
* chronic inflammatory disease
* rheumatoid arthritis
* pregnancy
* patients not able to give written consent
* patients with an implantable cardiac defibrillator or pacemaker
* patients which are sensitive to electromagnetic radiance

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-04-18 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Two Point Discrimination | 1 year
  Two Point Discrimination distal of the nerve lesion in mm
Semmes Weinstein Monofilament test | 1 year
  Palpable Monofilaments, measured in Newton
Pain/Discomfort | 1 year
  0=Hinders function 1=Disturbing 2=Moderate 3=None/minor
hyperesthesia | 1 year
  0=Hinders function 1=Disturbing 2=Moderate 3=None/minor

SECONDARY OUTCOMES:
Tinel Hoffmann sign | 1 year
  Progression of TH sign into the periphery
Sonography | 1 year
  sonography of the coaptation neuroma, measurement of the maximum diameter in mm
velocity of nerve conduction | 1 year
  Determination of velocity of nerve conduction
Medical Research Council Grading of Sensibility | 1 year
  Grading by the british medical research council. S0: No recovery of sensibility S1: Deep cutaneous pain sensibility S1+: superficial pain sensibility S2: superficial pain and some touch sensibility S2+: As in S2 but with overresponse S3: Pain and touch sensibility with over response, 2PD > 15mm S3+: As S3 but with imperfect recovery of 2PD (7-15mm) S4: Complete recovery

CONTACTS AND LOCATIONS:
Locations (2):
- Austria (2):
  - Meidling Trauma Hospital, Vienna
  - Lorenz Böhler Trauma Hospital, Vienna

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bosch G, Lin YL, van Schie HT, van De Lest CH, Barneveld A, van Weeren PR. Effect of extracorporeal shock wave therapy on the biochemical composition and metabolic activity of tenocytes in normal tendinous structures in ponies. Equine Vet J. 2007 May;39(3):226-31. doi: 10.2746/042516407x180408. PMID 17520973
- [Background] Corson MA, James NL, Latta SE, Nerem RM, Berk BC, Harrison DG. Phosphorylation of endothelial nitric oxide synthase in response to fluid shear stress. Circ Res. 1996 Nov;79(5):984-91. doi: 10.1161/01.res.79.5.984. PMID 8888690
- [Background] Fleming I, Bauersachs J, Fisslthaler B, Busse R. Ca2+-independent activation of the endothelial nitric oxide synthase in response to tyrosine phosphatase inhibitors and fluid shear stress. Circ Res. 1998 Apr 6;82(6):686-95. doi: 10.1161/01.res.82.6.686. PMID 9546377
- [Background] Fukumoto Y, Ito A, Uwatoku T, Matoba T, Kishi T, Tanaka H, Takeshita A, Sunagawa K, Shimokawa H. Extracorporeal cardiac shock wave therapy ameliorates myocardial ischemia in patients with severe coronary artery disease. Coron Artery Dis. 2006 Feb;17(1):63-70. doi: 10.1097/00019501-200602000-00011. PMID 16374144
- [Background] Hausdorf J, Sievers B, Schmitt-Sody M, Jansson V, Maier M, Mayer-Wagner S. Stimulation of bone growth factor synthesis in human osteoblasts and fibroblasts after extracorporeal shock wave application. Arch Orthop Trauma Surg. 2011 Mar;131(3):303-9. doi: 10.1007/s00402-010-1166-4. Epub 2010 Aug 22. PMID 20730589
- [Background] Martini L, Giavaresi G, Fini M, Torricelli P, de Pretto M, Schaden W, Giardino R. Effect of extracorporeal shock wave therapy on osteoblastlike cells. Clin Orthop Relat Res. 2003 Aug;(413):269-80. doi: 10.1097/01.blo.0000073344.50837.cd. PMID 12897619
- [Background] Moretti B, Notarnicola A, Garofalo R, Moretti L, Patella S, Marlinghaus E, Patella V. Shock waves in the treatment of stress fractures. Ultrasound Med Biol. 2009 Jun;35(6):1042-9. doi: 10.1016/j.ultrasmedbio.2008.12.002. Epub 2009 Feb 25. PMID 19243882
- [Background] Moretti B, Notarnicola A, Maggio G, Moretti L, Pascone M, Tafuri S, Patella V. The management of neuropathic ulcers of the foot in diabetes by shock wave therapy. BMC Musculoskelet Disord. 2009 May 27;10:54. doi: 10.1186/1471-2474-10-54. PMID 19473538
- [Background] Murata R, Nakagawa K, Ohtori S, Ochiai N, Arai M, Saisu T, Sasho T, Takahashi K, Moriya H. The effects of radial shock waves on gene transfer in rabbit chondrocytes in vitro. Osteoarthritis Cartilage. 2007 Nov;15(11):1275-82. doi: 10.1016/j.joca.2007.04.001. Epub 2007 May 29. PMID 17537650
- [Background] Nishida T, Shimokawa H, Oi K, Tatewaki H, Uwatoku T, Abe K, Matsumoto Y, Kajihara N, Eto M, Matsuda T, Yasui H, Takeshita A, Sunagawa K. Extracorporeal cardiac shock wave therapy markedly ameliorates ischemia-induced myocardial dysfunction in pigs in vivo. Circulation. 2004 Nov 9;110(19):3055-61. doi: 10.1161/01.CIR.0000148849.51177.97. Epub 2004 Nov 1. PMID 15520304
- [Background] Schaden W, Fischer A, Sailler A. Extracorporeal shock wave therapy of nonunion or delayed osseous union. Clin Orthop Relat Res. 2001 Jun;(387):90-4. doi: 10.1097/00003086-200106000-00012. PMID 11400900
- [Background] Schaden W, Thiele R, Kolpl C, Pusch M, Nissan A, Attinger CE, Maniscalco-Theberge ME, Peoples GE, Elster EA, Stojadinovic A. Shock wave therapy for acute and chronic soft tissue wounds: a feasibility study. J Surg Res. 2007 Nov;143(1):1-12. doi: 10.1016/j.jss.2007.01.009. Epub 2007 Sep 27. PMID 17904157
- [Background] Zimpfer D, Aharinejad S, Holfeld J, Thomas A, Dumfarth J, Rosenhek R, Czerny M, Schaden W, Gmeiner M, Wolner E, Grimm M. Direct epicardial shock wave therapy improves ventricular function and induces angiogenesis in ischemic heart failure. J Thorac Cardiovasc Surg. 2009 Apr;137(4):963-70. doi: 10.1016/j.jtcvs.2008.11.006. PMID 19327525